CLINICAL TRIAL: NCT03219710
Title: "Olanzapine for Prevention of Nausea and Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy (HEC): An Investigator Initiated, Randomized, Open-label Trial" (PRaCTiCE Trial: PRevention of ChemoTherapy Induced Emesis in Children)
Brief Title: "Olanzapine for Prevention of Chemotherapy Induced Nausea and Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy (HEC)"
Acronym: PRaCTiCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, RAMAVATH DEVENDRA NAIK, SENIOR RESIDENT, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IECPG-151/26.04.2017
Record Dates: First submitted 2017-05-10; First posted 2017-07-17 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Chemotherapy induced nausea and vomiting; olanzapine
MeSH Terms: conditions — Vomiting | interventions — Ondansetron; Dexamethasone; Aprepitant; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Patient on control group (ODA) with weight category of 15-40 kg will receive:
  D1-D3 Dexamethasone 3 mg/m2, ondansetron (0.15 mg/kg,), Aprepitant 80 mg;
  The patient on control group with weight category of > 40 kg will receive:
  D1- Dexamethasone 3 mg/m2 , ondansetron(0.15 mg/kg ), Aprepitant 125 mg; D2-D3 Dexamethasone 3mg/m2, ondansetron (0.15 mg/kg,), Aprepitant 80 mg
  Note: Aprepitant will be administered as single oral dose, dexamethasone and ondansetron will be administered q 8h (PO/IV)
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Aprepitant
- Arm B (Experimental): weight category of 15-40 kg will receive: D1-D3 Dexamethasone 3mg/m2, ondansetron (0.15 mg/kg,), Aprepitant 80 mg and olanzapine 0.14mg/kg (rounded off to nearest 2.5 mg) D4-olanzapine 0.14mg/kg (rounded off to nearest 2.5 mg)
  Weight category of > 40 kg in study group will receive:
  D1- Dexamethasone 3mg/m2, ondansetron (0.15 mg/kg, ), Aprepitant 125 mg; olanzapine 0.14mg/kg (rounded off to nearest 2.5 mg) D2-D3 Dexamethasone 3mg/m2, ondansetron (0.15 mg/kg,), Aprepitant 80 mg; olanzapine 0.14mg/kg (rounded off to nearest 2.5 mg) D4-olanzapine 0.14mg/kg (rounded off to nearest 2.5 mg) Note: Aprepitant & Olanzapine will be administered as single oral dose, dexamethasone and ondansetron will be administered q 8h (PO/IV)
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Aprepitant; Drug: Olanzapine

INTERVENTIONS:
Drug: Ondansetron — Ondansetron will be given at a dosage of 0.15mg/kg IV/PO q8h.
Drug: Dexamethasone — Dexamethasone will be given as 3mg/m2 IV/PO q8h.
Drug: Aprepitant — Aprepitant will be given as per the weight. weight (15-40kg) - Day1 to Day 3 - 80 mg PO weight (>40 kg) - Day 1 -125mg , Day 2 & Day 3 - 80 mg PO
Drug: Olanzapine — olanzapine will be given as 0.14mg/kg PO (rounded off to nearest 2.5 mg )
  Arms: Arm B

SUMMARY:
Chemotherapy induced nausea and vomiting (CINV) is one of the most distressing toxicities of cancer treatment. It can occur up to 90% in case of highly emetogenic chemotherapy (HEC) use. It is important to effectively manage CINV for a number of reasons. Acute phase vomiting can lead to vomiting in the delayed phase. It causes poor compliance with further therapy. Quality of life is compromised. It is easier to prevent nausea/vomiting than to treat it. Though strategies for prevention of CINV have been improved, it is still a significant problem. Newer drugs were explored and studied. The complete response rates were further increased with usage of olanzapine, an FDA approved antipsychotic, which blocks multiple neurotransmitters in the central nervous system.

Olanzapine has been studied in multiple randomized trials in adults for its safety and efficacy in prevention of CINV. Various RCTs have demonstrated the superiority of olanzapine for prevention of CINV in patients receiving highly and moderately emetogenic chemotherapy. Olanzapine has been approved for prevention of CINV in adults.

Unfortunately there are no large randomized trials demonstrating the efficacy of olanzapine for CINV prevention in children receiving HEC. The positive experience with olanzapine reported in adult oncology patients has prompted some pediatric clinicians to prescribe olanzapine for individual children receiving chemotherapy. Olanzapine is frequently used for the treatment of schizophrenia and bipolar disorder in children and adolescents. Though various studies have demonstrated safety of olanzapine in children, data regarding the efficacy of olanzapine in children and adolescents for prevention of CINV is limited. There are many small studies describing the safety and efficacy of olanzapine for prevention of CINV. However, there are no large randomized trials. Olanzapine is available in generic form and is not an expensive drug. Therefore we would like to conduct a randomized trial to look for the efficacy of olanzapine in pediatric population for prevention of CINV

DETAILED DESCRIPTION:
Children and adolescents registered with confirmed diagnosis of cancer will be assessed for eligibility criteria and enrolled in the study. Subjects will be randomized into study and control groups using table of random numbers generated by computer. Sequentially numbered, opaque, sealed envelopes will be used for concealed allocation. After randomization, subjects will be interviewed 1 hour prior 1st dose of chemotherapy. Subjects will receive the antiemetic drugs for four days as per the allotted arm. All doses will be administered under supervision and 30 minutes before chemotherapy. The data will be collected from each patient from day 1 to day5 from the last dose of chemotherapy. The details will contain different items dealing with demographic and clinical characteristic of the subjects. A Diary will be maintained for nausea and vomiting episodes. It will help in collecting data regarding nausea, vomiting along with some additional variables like chemotherapy related toxicities, requirement of any rescue medication. The subjects will be given the diary for symptom assessment on day 1 and it will be filled up under the supervision of the investigator on day 1 till completion of chemotherapy. The diary will be given to the subjects following the completion of chemotherapy to record all the events (incidence and severity of nausea, vomiting, requirement of rescue medication and other toxicities ) and will be contacted by phone or in person by the investigator. Edmonton's symptom assessment criterion will be used in the diary for assessing severity of nausea. The NCI's CTCAEv4.03 criterion will be used to assess the severity of vomiting and adverse events based on the data provided by the patient in the diary. Patients/attendants will be explained about the filling of the diary and will maintain it for recording of vomiting. A modified intention-to-treat population will be used for efficacy analysis. Proportion of patients with CR during acute phase, delayed phase and overall period will be compared between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age group 5-18 years with weight between ≥15 kg
* All subjects must have a confirmed diagnosis of malignancy
* European Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Scheduled to receive highly emetogenic chemotherapy as assessed using the Pediatric Oncology Group of Ontario Guideline for emetogenicity Classification
* Patients receiving first cycle of chemotherapy
* Children's caregiver who can understand Hindi or English and are willing to participate in the study (with written informed consent)

Exclusion Criteria:

* Have had treatment within 14 days prior to study enrollment with olanzapine or 30 days prior to study enrollment with another antipsychotic agent
* Planned to receive quinolone antibiotics while receiving olanzapine
* Have uncontrolled hypertension
* Receive other antipsychotic agents, amifostine, citalopram, CYP1A2 inducers or inhibitors
* Have a history of neuroleptic malignant syndrome, a seizure disorder, hypersensitivity to olanzapine.
* Children with known cardiac disease
* Are pregnant or breast-feeding
* Had received or will receive RT to abdomen or pelvis in the week prior to treatment
* Vomited in the 24 hours prior to study
* Previous exposure to HEC
* Abnormal lab values (ANC<1500/mm3, TLC<3000/mm3, Plt<100,000/mm3, AST/ALT> 2.5 times of ULN, bill>1.5 times of ULN, S.cr>1.5 times of ULN, patient on systemic steroids

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The number of patients with no episodes of vomiting as assessed by CTCAE v4.03 till 120 hours after highly emetogenic chemotherapy. | 120 hours after administration of chemotherapy.
  The number of patients achieving complete response as defined as, no episode of vomiting , assessed by CTCAE v.4.03 will be compared between the groups.
The number of patients with no episodes of vomiting as assessed by CTCAE v.03 till 24 hours after highly emetogenic chemotherapy. | Till 24 hours after administration of chemotherapy.
  The number of patients achieving complete response: defined as, no episode of vomiting , assessed by CTCAE v.4.03 will be compared between the groups.
The number of patients with no episodes of vomiting as assessed by CTCAE v4.03after 24 hours till 120 hours post highly emetogenic chemotherapy. | From 24 hours till 120 hours post administration of chemotherapy.
  The number of patients achieving complete response as defined as, no episode of vomiting , assessed by CTCAE v.4.03 will be compared between the groups.

SECONDARY OUTCOMES:
The number of patients with no episodes of nausea as assessed by "Edmonton symptom assessment scale" till 24 hours after highly emetogenic chemotherapy. | Till 24 hours after administration of chemotherapy.
  The no.of patients with no nausea, assessed by "Edmonton symptom assessment scale" during the study period will be compared between the groups
The number of patients with no episodes of nausea as assessed by "Edmonton symptom assessment scale" after 24 hours till 120 hours post highly emetogenic chemotherapy. | After 24 hours till 120 hours post administration of chemotherapy.
  The no.of patients with no nausea, assessed by "Edmonton symptom assessment scale" during the study period will be compared between the groups
The number of patients with no episodes of nausea as assessed by "Edmonton symptom assessment scale" till 120 hours post highly emetogenic chemotherapy. | Till 120 hours after administration of chemotherapy.
  The no.of patients with no nausea, assessed by "Edmonton symptom assessment scale" during the study period will be compared between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Bra Irch, Aiims, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naik RD, V S, Singh V, Pillai AS, Dhawan D, Bakhshi S. Olanzapine for Prevention of Vomiting in Children and Adolescents Receiving Highly Emetogenic Chemotherapy: Investigator-Initiated, Randomized, Open-Label Trial. J Clin Oncol. 2020 Nov 10;38(32):3785-3793. doi: 10.1200/JCO.20.00871. Epub 2020 Sep 15. PMID 32931400